CLINICAL TRIAL: NCT01332240
Title: External ValidatIon Trial of Aster: the Need for Surgical Staging After Echo-endoscopic Mediastinal Staging in Clinical N2/3 Lung Cancer
Brief Title: External ValidatIon Trial of ASTER Trial
Acronym: EVITA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EVITA001
Record Dates: First submitted 2011-04-05; First posted 2011-04-11 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-04

CONDITIONS: Stage III Lung Cancer
Keywords: staging; endosonography; lung cancer; stage III
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endosonography (Experimental): Endoscopic ultrasonography (EBUS-TBNA +/- EUS-FNA) for invasive mediastinal nodal staging
  Interventions: Procedure: Endoscopic ultrasonography

INTERVENTIONS:
Procedure: Endoscopic ultrasonography — in order to stage the mediastinum

SUMMARY:
As the use of endoscopic ultrasonography for mediastinal diagnosis and/or staging is widely spread in Belgium, the investigators aimed to determine the number of mediastinoscopies needed to detect one additional mediastinal lymph node invasion during routine clinical practice in the staging of potentially resectable clinical stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
Background : The observation made by the ASTER investigators might be criticized as all procedures were performed in highly experienced centers. To date, the number of mediastinoscopies needed to detect one additional N2/3 disease in the routine clinical practice of chest physician performing endosonography for mediastinal staging is unknown. The investigators therefore seek to answer whether a negative endosonography should routinely be followed by mediastinoscopy in day to day clinical practice.

Aim : As the use of endoscopic ultrasonography for mediastinal diagnosis and/or staging is widely spread in Belgium, the investigators aimed to determine the number of mediastinoscopies needed to detect one additional mediastinal lymph node invasion during routine clinical practice.

Setting : centers in Belgium with EBUS-TBNA and/or EUS-FNA experience in at least 20 patients agreed to participate and will include their patients.

Design : Prospective national observational multicenter study. All patients with clinical N2/3 disease based on CT and/or PET requiring invasive mediastinal staging will primarily undergo invasive mediastinal staging with endosonography (EBUS +/- EUS). A subsequent cervical mediastinoscopy will be performed in case no mediastinal lymph node involvement was found with endosonography. Local surgeons perform these procedures according to their institutional practice. Thoracotomy with mediastinal lymph node dissection will be the gold standard for invasive mediastinal staging, in case no mediastinal lymph node metastases were found during clinical staging including endosonography and mediastinoscopy.

Patients : The study will include 255 patients, based on the calculation of 15 consecutive patients in each participating center, in order to validate the ASTER data.

Primary endpoint : The number of mediastinoscopies needed to detect one additional N2/3.

Secondary endpoints : The number of mediastinal lymph nodes stations sampled with endosonography ; the median size of largest mediastinal lymph node sampled; characteristics of mediastinal nodal disease missed by endosonography.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with (suspected) NSCLC in whom invasive mediastinal staging is required based on presence of ACCP group B mediastinal lymph nodes and/or FDG-PET positive (visual interpretation of FDG uptake in mediastinal nodes as present) mediastinal lymph nodes (either ACCP group B or ACCP group D) in lymph node stations 2, 4, 7, 8 or 9 (see Appendix).
* Potentially operable and resectable disease.
* Radically treated previous extrathoracic malignancies are allowed whenever the extrathoracic malignancy is considered in remission, and a primary parenchymal lung tumour is present.
* Provision of a written informed consent.

Exclusion Criteria:

* Previous cervical mediastinoscopy.
* Uncorrected coagulopathy.
* Former treatment for a lung cancer.
* Patient unable to give a written informed consent.
* Absence of a primary parenchymal lung tumour.
* Distant metastases (cM1 disease) after routine clinical work-up.
* Clinical N2/3 disease only based on suspected mediastinal lymph nodes in stations 5 or 6.
* Patients belonging to ACCP groups A and C based on CT scan.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The number of mediastinoscopies needed to detect one additional N2/3 | 1 month
  Efficacy

SECONDARY OUTCOMES:
The number of mediastinal lymph nodes stations sampled with endosonography | 1 month
  Characteristics of nodal staging; the median size of largest mediastinal lymph node sampled; characteristics of mediastinal nodal disease missed by endosonography.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dooms, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Kurt Tournoy, Principal Investigator — University Hospital Ghent Belgium
Locations (18):
- Belgium (18):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Middelheim Ziekenhuis, Antwerp
  - Imelda ziekenhuis, Bonheiden
  - Sint-Jan Ziekenhuis Brugge, Bruges
  - Hopital Erasme Brussels, Brussels
  - Centre Hospitalier Universitaire de Charleroi, Charleroi
  - AZ Monica, Deurne
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Jesse Ziekenhuis, Hasselt
  - Univeristair Ziekenhuis Brussel, Jette
  - Center Hospitalier Jolimont, La Louvière
  - UCL, Mont-Godinne
  - Hopital Sainte-Elisabeth, Namur
  - Mariaziekenhuis, Overpelt
  - Heilig Hart Ziekenhuis, Roeselare
  - Sint-Elisabeth en Sint-Jozef ziekenhuis, Turnhout
  - Sint-Augustinus ziekenhuis, Wilrijk
  - UCL Saint-Luc, Woluwe